CLINICAL TRIAL: NCT01587521
Title: Prevalence of and Factors Associated With Metabolic Syndrome in Patients With Schizophrenia
Brief Title: Prevalence of and Factors Associated With Metabolic Syndrome in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Sirijit Suttajit, Assistant professor, Chiang Mai University
Other Study IDs: PSY-11-07-26A-12
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Metabolic Syndrome; Quality of Life; Depression
Keywords: Metabolic syndrome; Prevalence; Quality of life; Depression; Antipsychotics
MeSH Terms: conditions — Metabolic Syndrome; Depression

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with schizophrenia are more likely to have metabolic syndrome compared to general population. The criterion for metabolic syndrome in Asian people including: elevated waist circumference (male ≥ 90cm, female ≥ 80cm), elevated triglycerides ≥ 150mg/dL, reduced HDL cholesterol: male < 40mg/dL, female < 50mg/dL, elevated blood pressure: ≥ 130/85 mmHg, elevated fasting glucose: ≥ 100mg/dL. Several factors have been found to be associated with metabolic syndrome in schizophrenia, e.g. age, antipsychotic drugs, smoking, family history of metabolic disorder, stress, and quality of life.

However, little is known about the prevalence of and factors associated in Asian. This study aimed to:

1. Identify the prevalence of metabolic syndrome in patients with schizophrenia.
2. Identify the factors associated with metabolic syndrome in patients with schizophrenia.

DETAILED DESCRIPTION:
Patients with schizophrenia are more likely to have metabolic syndrome compared to general population. The criterion for metabolic syndrome in Asian people including: elevated waist circumference (male ≥ 90cm, female ≥ 80cm), elevated triglycerides ≥ 150mg/dL, reduced HDL cholesterol: male < 40mg/dL, female < 50mg/dL, elevated blood pressure: ≥ 130/85 mmHg, elevated fasting glucose: ≥ 100mg/dL. Several factors have been found to be associated with metabolic syndrome in schizophrenia, e.g. age, antipsychotic drugs, smoking, family history of metabolic disorder, stress, and quality of life.

However, little is known about the prevalence of and factors associated in Asian. This study aimed to:

1. Identify the prevalence of metabolic syndrome in patients with schizophrenia.
2. Identify the factors associated with metabolic syndrome in patients with schizophrenia.

Method This study is a cross-sectional study conducting at the Faculty of Medicine, Chiang Mai University. Eighty participants will be recruited with the inclusion criteria of having diagnosed with schizophrenia according to DSM-IV-TR and aged 18 years or over. The exclusion criterion is having organic brain syndrome.

Measurements PANSS CDSS WHOQOL-BREF-THAI

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-IV-TR
* Aged 18 years-old or over

Exclusion Criteria:

* Having organic brain syndromes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sirijit Suttajit, MD. MSc., Study Director — Chiang Mai University
Locations (1):
- Chiang Mai University, Chiang Mai, Chiang Mai, Thailand